CLINICAL TRIAL: NCT03214081
Title: Special Drug Use Surveillance of Takecab Tablets for "Maintenance Therapy of Reflux Esophagitis: Long-term Use"
Brief Title: Special Drug Use Surveillance of Vonoprazan for "Maintenance Therapy of Reflux Esophagitis: Long-term Use"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vonoprazan-5003; JapicCTI-163202 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vonoprazan 10 mg or 20 mg: Usually, for adults, 10 mg of vonoprazan administered orally once daily. If that dosing proved insufficient, the dosage may have been increased up to 20 mg once daily. Participants received vonoprazan as part of a routine medical care.
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: Takecab tablets; TAK-438

SUMMARY:
The purpose of this survey is to evaluate the safety and effectiveness of long-term administration of vonoprazan tablets when used as maintenance therapy for reflux esophagitis in routine clinical settings.

DETAILED DESCRIPTION:
The drug being tested in this survey is called vonoprazan. Vonoprazan is being tested to treat patients who have reflux esophagitis.

This survey will look at the safety and effectiveness of long-term administration of vonoprazan tablets when used as maintenance therapy for reflux esophagitis in routine clinical settings. The survey will enroll approximately 1000 participants.

- Vonoprazan 10 mg or 20 mg

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

- Participants who require maintenance therapy for relapsed/recurrent reflux esophagitis

Exclusion Criteria:

* Participants meeting the criteria of grade A to D according to the Los Angeles classification (Hoshihara's modification), by means of endoscopy at the initiation of maintenance therapy with vonoprazan tablets
* Participants with a previous history of hypersensitivity to ingredients in vonoprazan tablets
* Participants taking atazanavir sulfate or rilpivirine hydrochloride

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of participants with a diagnosis of reflux esophagitis and received dose of vonoprazan in the routine medical care.
Sampling Method: Probability Sample
Enrollment: 1237 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 122 investigative sites in Japan, from 01 March 2016 to 31 August 2018.
Pre-assignment Details: Participants with a historical diagnosis of reflux esophagitis were enrolled. Participants received vonoprazan as part of a routine medical care.
Period: Overall Study
Arm/Group | Vonoprazan 10 mg or 20 mg
Started | 1237
Completed | 1174
Not Completed | 63
Not completed — Case Report Forms Uncollected | 9
Not completed — Protocol Deviation | 54

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1174
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (13.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 683
  Male | 491
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 1174
Duration of Diagnosis of Reflux esophagitis [Mean (Standard Deviation); unit: Days] — Mean duration between start of study and first time of diagnosis of reflux esophagitis was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Days
    number analyzed (Participants) | 666
    (all) | 1109.5 (1449.98)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 1146
    Inpatient | 28
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported.
  Participants
    Had No Predisposition to Hypersensitivity | 1045
    Had Predisposition to Hypersensitivity | 72
    Unknown | 57
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 394
    Had Medical Complications | 780
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 727
    (all) | 157.86 (9.727)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 781
    (all) | 58.05 (12.985)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 725
    (all) | 23.17 (3.862)
Helicobacter Pylori Infection [Count of Participants; unit: Participants] — Number of participants with or without history of H. pylori infection was reported. "Negative" indicates the absence of H. pylori infection, "Positive" indicates presence of the infection.
  Participants
    Negative | 664
    Positive | 72
    Unknown | 438
Medical History of Esophageal Hiatal Hernia [Count of Participants; unit: Participants] — Number of participants with or without medical history of esophageal hiatal hernia was reported.
  Participants
    Had No Esophageal Hiatal Hernia | 591
    Had Esophageal Hiatal Hernia | 425
    Unknown | 158
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 563
  Current Smoker | 100
  Ex-Smoker | 181
  Unknown | 330
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 156
    No | 701
    Unknown | 317
Endoscopic Findings [Count of Participants; unit: Participants] — Endoscopic findings were assessed using the modified Los Angeles (LA) classification. The modified LA classification graded as follows- Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity; Grade A: non-confluent mucosal breaks <5 mm in length; Grade B: nonconfluent mucosal breaks ≥ 5mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >75% circumferential. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 1051
    Grade N | 130
    Grade M | 205
    Unassessed | 716
Prior Treatment with Acid Suppressants [Count of Participants; unit: Participants] — Number of participants who had or had not been treated with acid suppressants for reflux esophagitis was reported.
  Participants
    Had No Prior Treatment with Acid Suppressants | 214
    Had Prior Treatment with Acid Suppressants | 931
    Unknown | 29
Purpose of Acid Suppressants Treatment [Count of Participants; unit: Participants] — The purpose of treatment for those who received prior treatment with acid suppressants was reported. Population: Population Analysis Description: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 931
    Curative Therapy for Reflux Esophagitis | 325
    Maintenance Therapy for Reflux Esophagitis | 606

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1174
Percentage of Participants | 2.30

2. Secondary Outcome: Endoscopic Relapse Rate
Description: Endoscopic relapse rate was defined as a percentage of participants who met the criteria of Grade A to D in the modified Los Angeles (LA) classification. The modified LA classification graded endoscopic findings as follows- Grade N: normal mucosa; Grade M: minimal changes to the mucosa, such as erythema and/or whitish turbidity; Grade A: non-confluent mucosal breaks <5 mm in length; Grade B: nonconfluent mucosal breaks ≥ 5 mm in length; Grade C: confluent mucosal breaks <75% circumferential; Grade D: confluent mucosal breaks >=75% circumferential.
Time Frame: From the initiation of the maintenance therapy to Month 12 (or discontinuation of the therapy), up to 12 months
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 425
Percentage of Participants | 4.00 [2.35 to 6.33]

3. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Heartburn
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe heartburn at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available. Number analyzed is the number of participants who were evaluable at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 664
  Baseline: Mild | 368
  Baseline: Moderate | 270
  Baseline: Severe | 26
  Month 6: number analyzed (Participants) | 155
  Month 6: Mild | 136
  Month 6: Moderate | 17
  Month 6: Severe | 2
  Month 12: number analyzed (Participants) | 91
  Month 12: Mild | 84
  Month 12: Moderate | 7
  Month 12: Severe | 0

4. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Acid Reflux
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe acid reflux at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 471
  Baseline: Mild | 292
  Baseline: Moderate | 159
  Baseline: Severe | 20
  Month 6: number analyzed (Participants) | 112
  Month 6: Mild | 94
  Month 6: Moderate | 16
  Month 6: Severe | 2
  Month 12: number analyzed (Participants) | 63
  Month 12: Mild | 52
  Month 12: Moderate | 11
  Month 12: Severe | 0

5. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Postprandial Fullness
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe postprandial fullness at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 283
  Baseline: Mild | 196
  Baseline: Moderate | 77
  Baseline: Severe | 10
  Month 6: number analyzed (Participants) | 70
  Month 6: Mild | 61
  Month 6: Moderate | 7
  Month 6: Severe | 2
  Month 12: number analyzed (Participants) | 45
  Month 12: Mild | 40
  Month 12: Moderate | 5
  Month 12: Severe | 0

6. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Early Satiation
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe early satiation at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 108
  Baseline: Mild | 80
  Baseline: Moderate | 23
  Baseline: Severe | 5
  Month 6: number analyzed (Participants) | 38
  Month 6: Mild | 29
  Month 6: Moderate | 7
  Month 6: Severe | 2
  Month 12: number analyzed (Participants) | 25
  Month 12: Mild | 21
  Month 12: Moderate | 4
  Month 12: Severe | 0

7. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Epigastric Pain
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe epigastric pain at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 232
  Baseline: Mild | 167
  Baseline: Moderate | 52
  Baseline: Severe | 13
  Month 6: number analyzed (Participants) | 69
  Month 6: Mild | 63
  Month 6: Moderate | 6
  Month 6: Severe | 0
  Month 12: number analyzed (Participants) | 44
  Month 12: Mild | 40
  Month 12: Moderate | 4
  Month 12: Severe | 0

8. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Epigastric Burning
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe epigastric burning at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 158
  Baseline: Mild | 97
  Baseline: Moderate | 49
  Baseline: Severe | 12
  Month 6: number analyzed (Participants) | 32
  Month 6: Mild | 28
  Month 6: Moderate | 3
  Month 6: Severe | 1
  Month 12: number analyzed (Participants) | 10
  Month 12: Mild | 9
  Month 12: Moderate | 1
  Month 12: Severe | 0

9. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Abdominal Bloating
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe abdominal bloating at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 127
  Baseline: Mild | 91
  Baseline: Moderate | 31
  Baseline: Severe | 5
  Month 6: number analyzed (Participants) | 48
  Month 6: Mild | 40
  Month 6: Moderate | 5
  Month 6: Severe | 3
  Month 12: number analyzed (Participants) | 33
  Month 12: Mild | 28
  Month 12: Moderate | 5
  Month 12: Severe | 0

10. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Nausea/Vomiting
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe nausea/vomiting at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 96
  Baseline: Mild | 69
  Baseline: Moderate | 25
  Baseline: Severe | 2
  Month 6: number analyzed (Participants) | 38
  Month 6: Mild | 28
  Month 6: Moderate | 9
  Month 6: Severe | 1
  Month 12: number analyzed (Participants) | 21
  Month 12: Mild | 20
  Month 12: Moderate | 1
  Month 12: Severe | 0

11. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Belching
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe belching at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 206
  Baseline: Mild | 138
  Baseline: Moderate | 60
  Baseline: Severe | 8
  Month 6: number analyzed (Participants) | 71
  Month 6: Mild | 62
  Month 6: Moderate | 7
  Month 6: Severe | 2
  Month 12: number analyzed (Participants) | 57
  Month 12: Mild | 51
  Month 12: Moderate | 6
  Month 12: Severe | 0

12. Secondary Outcome: Number of Participants With Recorded Severity of Subjective Symptoms of Anorexia
Description: Presence or absence and severity of subjective symptoms were collected from participants during medical interviews of each visit as none (asymptomatic), mild (occasionally or slightly symptomatic), moderate (considerably symptomatic), severe (unendurably symptomatic), and unknown. Number of participants who had mild, moderate, or severe anorexia at each time points were reported.
Time Frame: Baseline, Month 6 and at Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg or 20 mg
Number analyzed (Participants) | 1141
Participants
  Baseline: number analyzed (Participants) | 105
  Baseline: Mild | 67
  Baseline: Moderate | 33
  Baseline: Severe | 5
  Month 6: number analyzed (Participants) | 46
  Month 6: Mild | 35
  Month 6: Moderate | 9
  Month 6: Severe | 2
  Month 12: number analyzed (Participants) | 19
  Month 12: Mild | 15
  Month 12: Moderate | 4
  Month 12: Severe | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Vonoprazan 10 mg or 20 mg
All-Cause Mortality (participants affected / at risk) | 7/1174
Serious Adverse Events (participants affected / at risk) | 15/1174
Other Adverse Events (participants affected / at risk) | 11/1174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg or 20 mg (N=1174)
Pneumonia (Infections and infestations) | 2
Peritonitis bacterial (Infections and infestations) | 1
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelopathy (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Angina unstable (Cardiac disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Death (General disorders) | 1 — The event had a causal relationship with a complication of ureteral cancer, and the causality of the event was "not related" to vonoprazan.
Platelet count decreased (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg or 20 mg (N=1174)
Diarrhoea (Gastrointestinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03214081/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03214081/SAP_001.pdf